CLINICAL TRIAL: NCT06542380
Title: TAVI PACER: A Two-step Risk Score for Prediction of Permanent Pacemaker Implantation After TAVI.
Acronym: TAVI PACER
Status: Completed | Type: Observational
Sponsor: German Heart Institute (Other)
Responsible Party: Principal Investigator, Julia Lueg, Principal Investigator, German Heart Institute
Other Study IDs: DRKS00024852
Record Dates: First submitted 2024-07-19; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-07

CONDITIONS: Pacemaker; TAVI; Risk Score
Keywords: Transcatheter aortic valve replacement; Aortic stenosis; Pacemaker implantation; Risk Score; Electrocardiogram; Risk Stratification
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing TAVI at DHZC 2019-2021
  Interventions: Device: TAVI, pacemaker

INTERVENTIONS:
Device: TAVI, pacemaker — Retrospective analysis of need for pacemaker implantation after TAVI

SUMMARY:
The need for permanent pacemaker implantation (PPMI) remains one of the most frequent complications after transcatheter aortic valve implantation (TAVI). This study aimed to develop a novel, two-step risk score to predict PPMI probability after TAVI and to implement it into a user-friendly website. Our risk score addresses the gap in existing data on current prosthesis generations and provides a new and clinically motivated approach to calculating the risk for PPMI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing TAVI at Deutsches Herzzentrum der Charité between January 2019 and December 2020

Exclusion Criteria:

* previous device implantation
* valve-in-valve procedure
* patients who had received an ALLEGRATM valve (NVT AG, Morges, Switzerland), a LOTUS EdgeTM valve (Boston, Scientific, Natick, Massachusetts), or a CENTERATM valve (Edwards Lifesciences, Irvine, California)

Ages: 51 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Given the retrospective nature of the study, all patients who had undergone TAVI at the DHZC were included, with the exception of those meeting the exclusion criteria mentioned above. Consequently, the study population is primarily comprised of individuals aged 75 years and above, with a balanced gender distribution.
  Following current guidelines, every patient undergoing TAVI received an initial assessment by a multidisciplinary heart team.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-06-28 (Actual)

PRIMARY OUTCOMES:
Pacemaker Implantation | 30 days after TAVI
  Rate of pacemaker implantation up to 30 days after TAVI according to current guidelines

CONTACTS AND LOCATIONS:
Overall Officials: Henryk Dreger, Professor, Principal Investigator — German Heart Institute
Locations (1):
- Deutsches Herzzentrum der Charité, Mitte, State of Berlin, Germany